CLINICAL TRIAL: NCT04456101
Title: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Brief Title: Study on the Recovery of Pulmonary Function, Chest CT, Airway Microbiota, Hematologic, and Immune & Inflammatory Conditions in COVID-19 Rehabilitation Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Department of Respiratory and Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: NCIP03
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: healthy individuals without COVID-19
- Severe/Critical COVID-19 rehabilitation group: ①Individuals recovering from Severe/Critical COVID-19
- mild/moderate COVID-19 rehabilitation group: Individuals recovering from mild/moderate COVID-19
- asymptomatic COVID-19 rehabilitation group: Asymptomatic COVID-19 individuals with laboratory test for SRARS-COV2 turning negative

SUMMARY:
The intent of this study was to examine the health status of individuals who had been confirmed with COVID-19 in the year after their recovery. Parameters studied included serum levels of SARS coronavirus 2 (SARS-CoV 2) IgG antibody, SARS-CoV-2 nucleic acid test, hematology indicators (blood routine, liver function, kidney function, myocardial enzymes, coagulation function, etc), lung function test, imaging data and airway microbiota data. In addition, we explored the systematic Immune & Inflammation in some of the individuals recovering from COVID-19.

DETAILED DESCRIPTION:
About 20% of COVID-19 developed into a critical illness and about 2% died. The global epidemic continues to develop, but some patients in China have entered the rehabilitation period, which is accompanied by a large number of respiratory symptoms and pulmonary fibrosis, bringing serious harm to the country. Therefore, early accurate detection and prediction of the development trend of patients in rehabilitation period and targeted treatment measures for corresponding patients are the key to the success of COVID-19 rehabilitation period. It will play a key role in the stratified management of the post-epidemic situation, which is crucial to improve the quality of life of COVID-19 patients. We aim to explore the clinical characteristics of rehabilitation patients by detecting some indicators of patients in rehabilitation period, including serum IgG and IgM antibody of SARS-CoV 2, SARS-CoV-2 nucleic acid, hematology indicators (blood routine, liver function, kidney function, myocardial enzymes, coagulation function, etc), pulmonary function, chest CT imaging, systematic Immune & Inflammation states.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals recovering from COVID-19, or asymptomatic COVID-19 patients with laboratory test for SRARS-COV2 turning negative, or healthy volunteers without COVID-19.
2. The age range is 18-80 years.
3. Subjects or their family members agree to participate in the study and sign informed consent.
4. The previously diagnosed individuals have been cured for about 1 month.

Exclusion Criteria:

1. Woman who is breastfeeding, pregnant, or preparing to become pregnant.
2. Patients with cognitive impairment or poor compliance as determined by the investigator.
3. Participants in other clinical trials.
4. Subjects who were not suitable for clinical trials determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Covid-19 rehabilitation was the experimental group, and the healthy control group was the conventional control group
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function | an average of 1 to 3 months after recovery
  Forced vital capacity (FVC), forced expiratory volume in one second (FEV1) for lung volume, peak expiratory flow (PEF) for velocity, carbon monoxide diffusion capacity (DLCO) for pulmonary diffusion function.
Chest CT | an average of 1 to 3 months after recovery
  Percentage of lungs that contain reticular patterns, Percentage of lungs that contain pure ground-glass opacification, Percentage of lungs that contain honeycombing, Percentage of lungs that contain traction bronchiectasis, Percentage of lungs that contain strip-like consolidation.
Changes in hematology | an average of 1 to 3 months after recovery
  blood routine indexes included leucocytes(×109/L), neutrophils(×109/L), lymphocytes(×109/L), monocytes(×109/L), eosinophils(×109/L), platelets(×109/L). Biochemical and coagulation function indicators included total protein(umol/L), creatinine (umol/L), uric acid (umol/L), lactic dehydrogenase(U/L), C-reactive protein (mg/L), aspartate aminotransferase (U/L), glutamic-pyruvic transaminase (U/L), D-dimer,(ug/L), fibrinogen(g/L), Active part thrombin time (APTT), prothrombin time (PT), thrombin time (TT) and troponin (TNI).
Changes in immune and inflammatory states | an average of 1 to 3 months after recovery
  Immune cells and related cell factors included CD8+T cell(×109/L), CD4+T cell(×109/L), bone marrow derived suppressor cells(×109/L), regulatory T cells(×109/L), natural killer cell(×109/L), dendritic cell(×109/L), macrophages(×109/L), interleukin-4(IL-4)ug/L, IL-2 ug/L, IL-17 ug/L, IL-15 ug/L, IL-16 ug/L, IL-1 ug/L, IL-6 ug/L, IL-10 ug/L, tumor necrosis factor ug/L, interferon gamma ug/L, eotaxin-3 ug/L, eotaxin ug/L.
St. George's Respiratory Questionnaire(SGRQ) | an average of 1 to 3 months after recovery
  St. George's Respiratory Questionnaire total score(0-3989.4), St. George's Respiratory Questionnaire symptoms score(0-662.5); St. George's Respiratory Questionnaire impacts score(0-2117.8); St. George's Respiratory Questionnaire activity score(0-1209.1). The higher the score, the worse the lung.
Modified British medical research council (mMRC) | an average of 1 to 3 months after recovery
  mMRC only reflects symptom of dyspnea. A score of 0-1 is considered as fewer symptom, and ≥2 is considered as more symptom.
COPD Assessment test (CAT) | an average of 1 to 3 months after recovery
  CAT score was a comprehensive symptom score ranging from 0 to 40 points. The higher the score, the worse the lung.
Airway Microbiota | an average of 1 to 3 months after recovery
  Airway Microbiota of exhaled breath condensate in individuals were detected.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jin, professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No